CLINICAL TRIAL: NCT00462852
Title: A Phase II Randomized Study of Chemo-Anticoagulation (Gemcitabine-Dalteparin) Versus Chemotherapy Alone (Gemcitabine) for Locally Advanced and Metastatic Pancreatic Adenocarcinoma [FRAGEM]
Brief Title: Gemcitabine With or Without Dalteparin in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PRH-HCTU-FRAGEM; CDR0000540180 (Registry Identifier: PDQ (Physician Data Query)); PRH-HCTU-FRAGEM-V-12.1; CTA-MF8000/13558; EU-20721; LILLY-PRH-HCTU-FRAGEM; ISRCTN76464767
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer; Thromboembolism
Keywords: thromboembolism; stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism | interventions — Dalteparin; Gemcitabine

INTERVENTIONS:
Drug: dalteparin
Drug: gemcitabine hydrochloride
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Anticoagulants, such as dalteparin, may help prevent blood clots from forming in patients being treated with gemcitabine for pancreatic cancer.

PURPOSE: This randomized phase II trial is studying how well gemcitabine works with or without dalteparin in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of venous thromboembolism in patients with locally advanced or metastatic pancreatic cancer treated with gemcitabine hydrochloride and dalteparin versus gemcitabine hydrochloride alone.

Secondary

* Compare the survival benefit, in terms of increased (from 70% to 85%) survival at 12 weeks, of patients treated with these regimens.
* Compare the toxicity of these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the time to disease progression in patients treated with these regimens.
* Determine the effect of gemcitabine hydrochloride and dalteparin on serological markers of thromboangiogenesis.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to disease progression (locally advanced vs metastatic) and Karnofsky performance status (≥ 80% vs < 80%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 1-7 and 9-11.
* Arm II: Patients receive low molecular weight dalteparin subcutaneously once daily in weeks 1-12. Patients also receive gemcitabine hydrochloride as in arm I.

Blood samples are acquired at baseline for analysis of circulating tissue factor and vascular endothelial growth factor.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or locally advanced adenocarcinoma of the pancreas

  * Patients with clinical 'high probability' of pancreatic cancer and biopsy suggestive but not diagnostic of pancreatic cancer may be eligible based on review by the principal investigator
* Measurable or evaluable disease
* No clinical evidence of active venous thromboembolism

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 60-100% OR WHO PS 0-2
* Life expectancy > 12 weeks
* Absolute neutrophil count > 2,000/mm³
* WBC > 3,000/mm³
* Platelet count > 100,000/mm³
* Creatinine clearance > 50 mL/min
* INR ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN (stent allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No cerebrovascular accident within the past 6 months
* No obvious contraindication to anticoagulation, including the following:

  * Bleeding diathesis
  * Active peptic ulcer
  * Ulcerating cancer into duodenum
* No history of other advanced malignancy
* No gross hematuria
* No melaena or gross evidence of gastrointestinal bleeding (other than piles)
* No requirement for a central line
* No other significant medial or psychiatric illness that, in the opinion of the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior gemcitabine hydrochloride-containing treatment
* No other concurrent cytotoxic chemotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids), or experimental medications
* No other concurrent specific anticancer therapy as a result of disease progression
* No concurrent caval filter device
* No other concurrent anticoagulants for venous thromboembolism or other reasons (e.g., atrial fibrillation)
* No concurrent acetylsalicylic acid (> 75 mg) as an antiplatelet drug for a preexisting cardiovascular condition
* No concurrent clopidogrel bisulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-04; Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism reduction

SECONDARY OUTCOMES:
Early survival benefit
Toxicity
Overall survival
Time to disease progression
Effect of drug combination on serological markers of thromboangiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Maraveyas, Study Chair — Hull University Teaching Hospitals NHS Trust
Locations (8):
- United Kingdom (8):
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Saint Bartholomew's Hospital, London, England
  - St. George's Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Nottingham City Hospital, Nottingham, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Maraveyas A, Waters J, Roy R, Fyfe D, Propper D, Lofts F, Sgouros J, Gardiner E, Wedgwood K, Ettelaie C, Bozas G. Gemcitabine versus gemcitabine plus dalteparin thromboprophylaxis in pancreatic cancer. Eur J Cancer. 2012 Jun;48(9):1283-92. doi: 10.1016/j.ejca.2011.10.017. Epub 2011 Nov 17. PMID 22100906